CLINICAL TRIAL: NCT00938847
Title: Bone Marrow Derived Mononuclear Cells For Myocardial Regeneration in Early Left Ventricular Dysfunction After Acute Myocardial Infarction And Successful Percutaneous Coronary Intervention
Brief Title: Bone Marrow Derived Mononuclear Cells For Myocardial Regeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asklepios proresearch (Industry)
Collaborators: Cordis US Corp. (Industry)
Responsible Party: Prof. Dr. med. Karl-Heinz Kuck, Asklepios Klinik St. Georg, Departement of Cardiology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 996; 2005-003629-19; 2508
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Left Ventricular Dysfunction
Keywords: left ventricular dysfunction; myocardial infarction; left ventricular dysfunction (LVDF) after acute myocardial infarction
MeSH Terms: conditions — Ventricular Dysfunction, Left; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PCI — Stent implantation after acute myocardial infarction

SUMMARY:
Evaluative pilot study for safety and feasibility with administration of autologous bone bone marrow derived mononuclear cells by endoventricular catheter into the normal border zone fo the ischemic lesion.

ELIGIBILITY:
Inclusion Criteria:

* LVEF <40%
* PCI at latest 6 hours after infarction
* BMI >20 kg/m² and <30 kg/m²

Exclusion Criteria:

* PCI elder than 14 days
* relevant valvular disease
* left ventricular dysfunction caused by other reasons than ischemic cardiomyopathy
* history of stroke, chronic atrial fibrillation, multivessel disease, thromboembolic event
* scheduled for CABG
* DM Type 1 & extensive hypercholesterinemia
* pacemaker
* systemic disease
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-02; Primary Completion 2007-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Demonstration of safety and feasibility of BM-MNC treatment. Investigation of the suitability of endocardial left ventricular electromechanical mapping (LVEMM) with NOGA as endpoint for myocardial regeneration. | 12 months

SECONDARY OUTCOMES:
Collection of first evidence on the best type and time points for the determination of myocardial regeneration by NOGA and other parameters. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, Prof. Dr. med., Principal Investigator — Asklepios Klinik St. Georg, Departement of Cardiology
Locations (1):
- Asklepios Klinik St. Georg, Departement of Cardiology, Hamburg, Germany